CLINICAL TRIAL: NCT01964053
Title: Promoting Self-management Through Adherence Among Heart Failure Patients
Brief Title: Self-management Adherence in Heart Failure Patients
Acronym: PATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0228-13-EP
Record Dates: First submitted 2013-10-10; First posted 2013-10-17 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
Keywords: Self-management adherence; post acute care; critical access hospitals; patient activation; hospital readmission
MeSH Terms: conditions — Heart Failure; Patient Participation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PATCH Intervention (Experimental): The intervention group will receive usual care and the PATCH intervention. The intervention is comprised of two phases in which the in-hospital discharge education session is followed by 12 weeks of post-discharge education sessions delivered by telephone. The focus of this study is to test the mechanism of the proposed patient activation intervention on HF self-management adherence and associated health outcomes.
  Interventions: Behavioral: PATCH intervention
- Usual Care (Active Comparator): The usual care group will receive standardized discharge written information and scheduled doctor appointments. Standardized discharge instruction, as recommended by CMS and the Joint Commission, includes: activity level, diet, discharge medications, follow-up doctor appointment, weight monitoring, and what to do if symptoms worsen. No further follow-ups are routinely done by the hospital and patients are told to see their primary care provider if problems occur.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: PATCH intervention — The intervention group will receive usual care and the PATCH intervention. The intervention is comprised of two phases in which the in-hospital discharge education session is followed by 12 weeks of post-discharge education sessions delivered by telephone. The focus of this study is to test the mechanism of the proposed patient activation intervention on HF self-management adherence and associated health outcomes.
  Arms: PATCH Intervention
Behavioral: Usual care — Usual care refers to the standardized discharge written information and scheduled doctor appointments. Standardized discharge instruction, as recommended by CMS and the Joint Commission, includes: activity level, diet, discharge medications, follow-up doctor appointment, weight monitoring, and what to do if symptoms worsen.113 No further follow-ups are routinely done by the hospital and patients are told to see their primary care provider if problems occur.
  Arms: Usual Care

SUMMARY:
Non-adherence to self-management behaviors is prevalent and accounts for hospital readmissions in heart failure (HF) patients 65 years of age and older. The mechanism to activate and engage HF patients in managing their own care is uncertain. Yet post-acute care service that is vital to improve HF patients' self-management adherence and HF outcomes is suboptimal in rural hospitals (primarily critical access hospitals). The investigators central hypothesis is that patients with higher activation level will have significantly better self-management adherence. This study will test whether Patient AcTivated Care at Home (PATCH) will improve self-management adherence and health outcome (reduced hospital readmissions), as well as the feasibility to translate the research findings to a home based post-acute care service in rural communities.

DETAILED DESCRIPTION:
Heart failure (HF) is among the most prevalent chronic conditions and leading cause of hospital readmission in adults 65 years of age and older. HF patients discharged from rural critical access hospitals (CAHs) had higher 30-day readmission rates compared to patients discharged from urban hospitals. Adhering to recommended self-management behaviors improves HF patients' health outcomes and reduces readmissions; however, the prevalence of adherence is low in HF patients. In rural communities, low adherence can be attributed to the fact that rural HF patients received less information about managing their chronic condition based on the investigators preliminary study. Previous studies reported inconsistent findings regarding the effectiveness of interventions designed to improve self-management adherence. The feasibility of these interventions in rural settings is unknown. Therefore, innovative programs are needed to identify the intervention to enhance self-management adherence in HF patients living in rural communities. The purpose of this prospective, two-group, repeated measures, randomized control trial is to test the efficacy and feasibility of a 12-week activation-enhancing intervention (Patient AcTivated Care at Home [PATCH]) on self-management adherence and health outcome (readmission rates) in HF patients discharged from rural hospitals (critical access hospitals). A sample size of 96 subjects with heart failure will be recruited over 14 month period. Both intervention and control groups will receive usual care. The intervention group will additionally receive 2-phase PATCH intervention: the in-hospital discharge education session (Phase I) and 12-week post-discharge education sessions delivered by telephone (Phase II). The tailored strategies are developed to activate patients engaging in self-management behaviors based on their baseline activation level. The investigators central hypothesis, based upon their preliminary data, is that patients with higher activation level will have significantly better self-management adherence. The investigators will test their hypothesis with the following Specific Aims: To evaluate the effects of the patient activation intervention on self-management adherence (Aim 1) and hospital readmissions (Aim 2) over time. To evaluate the mechanism of the patient activation intervention (Aim 3). To evaluate the feasibility of the PATCH intervention (Aim 4). The PATCH intervention is innovative because: 1) it translates patient activation theory into intervention strategies to improve self-management in a vulnerable population (rural heart failure patients living in rural community), 2) it tests the mechanism of patient activation on self-management adherence; 3) it uses the rural nursing theory to guide developing a sustainable intervention program in rural communities; and 4) it evaluates a biomarker collected by a single urine test as the indicator of self-management adherence in HF patients. This study will impact the management of heart failure by adding knowledge about the mechanism to improve self-management adherence in heart failure patient living in rural communities. Long term adherence to the recommended self-management behaviors is the foundation to realize health benefit and reduce burden on patients, their family and the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* have HF as one of their discharge diagnoses;
* have New York Heart Association (NYHA) class II to IV symptoms or have NYHA class I symptoms
* have had at least one other HF-related hospitalization or emergency department visit in the previous year;
* are discharged to home;
* pass a mini-cog screen
* understand English;
* have access to a phone.

Exclusion Criteria:

* Have scheduled procedures and/or surgeries during hospitalization;
* Have depressive symptoms (receive a score of 3 or above on the Patient Health Questionnaire-2 (PHQ-2) have documented medical diagnosis or diagnostic evidence of liver cirrhosis;
* Have renal failure (serum creatinine greater than 2.0mg/dl)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in self-management adherence at 3 and 6 months | 3 and 6 months following intervention
  Primary outcome of self-management adherence refers to the adherence to self-care behaviors

SECONDARY OUTCOMES:
Change from Baseline in re-hospitalization rate at 30-day, 3 and 6 months | 30 day after intervention
  Evaluate the immediate and extended effects of the patient activation intervention on the re-hospitalization rate in heart failure patients

CONTACTS AND LOCATIONS:
Overall Officials: Lufei Young, PhD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Beatrice Community Hospital & Health Center, Beatrice, Nebraska
  - Jefferson Community Health Center, Fairbury, Nebraska

REFERENCES:
- [Derived] Young L, Hertzog M, Barnason S. Effects of a home-based activation intervention on self-management adherence and readmission in rural heart failure patients: the PATCH randomized controlled trial. BMC Cardiovasc Disord. 2016 Sep 8;16(1):176. doi: 10.1186/s12872-016-0339-7. PMID 27608624
- [Derived] Young L, Barnason S, Do V. Promoting self-management through adherence among heart failure patients discharged from rural hospitals: a study protocol. F1000Res. 2014 Dec 30;3:317. doi: 10.12688/f1000research.5998.2. eCollection 2014. PMID 25844160